CLINICAL TRIAL: NCT06919341
Title: RESTI Registry: Spanish Registry of Primary Immune Thrombocytopenia and Other Immune Thrombocytopenia
Acronym: RESTI
Status: Recruiting | Type: Observational
Sponsor: Fundación Española de Hematología y Hemoterapía (Other)
Responsible Party: Sponsor
Other Study IDs: RESTI
Record Dates: First submitted 2025-03-29; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: ITP - Immune Thrombocytopenia; Primary Immune Thrombocytopenia (ITP)
Keywords: ITP; PTI; Trombocitopenia inmune primaria; Primary Inmune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Primary immune thrombocytopenia (PIT), previously referred to as idiopathic thrombocytopenic purpura, is an acquired disease characterized by accelerated platelet destruction and deficient platelet production by megakaryocytes.

Although the existence of PIT has been known for decades, there is no consensus on its triggering mechanisms. On the other hand, this disease presents a very heterogeneous patient profile, both in its characteristics and treatments. In this sense, the diagnosis is still made by excluding other causes of thrombocytopenia.

There is insufficient epidemiological data on the disease, a fact that is especially evident in our country. We have no data on the incidence or prevalence of this pathology in Spain.

For all these reasons, this epidemiological study has been designed to increase the available knowledge about this disease and the detailed characterization of the population of patients with ITP in Spain.

The main objective of this study is to describe the clinical, analytical and treatment characteristics of primary immune thrombocytopenia and other immune thrombocytopenia.

The study is an epidemiological, ambispective, multicenter study carried out in hospitals in Spain.

Information will be collected on the disease under study, as well as on the treatments received, using the patient's clinical history as a source document.

ELIGIBILITY:
Inclusion Criteria:

* Children as young as 2 months of age and adults in follow-up since 2015 (irrespective of date of diagnosis) with the diagnostic presumption of PIT or other thrombocytopenia of probable immune origin defined as a platelet count < 100 x 109/L.
* Patients who have given written informed consent. In the case of deceased patients, the data will be included in the registry and the investigator will record the impossibility of collecting patient's informed consent form due to death. Only patients deceased after December 31 2015, will be included

Exclusion Criteria:

* Patients who, at the investigator's discretion, do not meet the conditions for inclusion in the study

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with the diagnostic presumption of PIT or other thrombocytopenia of probable immune origin defined as a platelet count < 100 x 109/L.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Description of the clinical and analytical features of PIT and other immune thrombocytopenias. | From enrollment

SECONDARY OUTCOMES:
Comparison with published historical ITP data | From enrollment
Definition of therapeutic strategies and most common treatments in ITP | From enrollment
Evaluation of response to first-line treatment | From enrollment
Evaluation of response to subsequent treatments | From enrollment

CONTACTS AND LOCATIONS:
Locations (36):
- Spain (36):
  - Complexo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital Del Mar, Barcelona, Barcelona
  - Hospital Vall d'Hebron (, Barcelona, Barcelona
  - Hospital Universitario Mutua Terrassa, Terrassa, Barcelona
  - Hospital de Basurto, Bilbao, Biskaia
  - Hospital Sierrallana, Torrelavega, Cantabria
  - Hospital de La Plana, Castellon, Castellón
  - Hospital Universitario Punta de Europa, Algeciras, Cádiz
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Universitario Reina Sofia de Córdoba, Córdoba, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Juan Ramón Jimenez, Huelva, Huelva
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario Arnau de Vilanova, Lleida, Lérida
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario 12 octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Costa del Sol, Marbella, Málaga
  - Hospital Universitario Regional de Málaga, Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital materno infantil de Málaga, Málaga, Málaga
  - Hospital de la Serranía de Ronda, Ronda, Málaga
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital de la Merced, Osuna, Sevilla
  - Hospital Universitario Virgen de la Macarena, Seville, Sevilla
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No